CLINICAL TRIAL: NCT02136758
Title: Cardiovascular Risk Clinic
Acronym: CRC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding cut due to government sequestration
Sponsor: Windber Research Institute (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-07; W81XWH-10-2-0080 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2014-05-08; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Disease; Coronary Artery Disease; Hypertension; Diabetes; Obesity
Keywords: lifestyle modification; diet; exercise; cardiovascular disease; gene expression; obesity
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Hypertension; Diabetes Mellitus; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle modification (Experimental): The intervention group participated in individualized therapeutic lifestyle plans to reduce cardiovascular risk. Participants were introduced to factors contributing to cardiovascular disease and met individually with a registered dietitian, exercise physiologist, stress management instructor, and psychologist to learn effective strategies for integrating healthy changes into their current lifestyle.
  Interventions: Behavioral: CRC lifestyle modification program
- Usual care controls (No Intervention): Control group received standard care from their primary physicians, but did not participate in any component of the lifestyle program or receive any information, advice, or counseling regarding healthy lifestyle behaviors.

INTERVENTIONS:
Behavioral: CRC lifestyle modification program — Intervention group enrolled in lifestyle program in which they developed individualized therapeutic lifestyle plans to reduce cardiovascular risk.
  Arms: Lifestyle modification

SUMMARY:
This study was a prospective, randomized trial designed to investigate the efficacy of moderate lifestyle modification for improving the clinical status of patients with coronary artery disease or patients with risk factors that promote coronary artery disease.

DETAILED DESCRIPTION:
The main hypothesis to be tested in the Cardiovascular Risk Clinic was: Can individualized therapeutic lifestyle plans in conjunction with molecular analysis lead to informative assessments of disease risk that can reduce risk factors for diabetes and cardiovascular disease.

Our main objectives were:

A. To investigate the effect of lifestyle modification on: (1) physiological measurements of coronary artery disease (CAD) including carotid intima-media thickness (CIMT), exercise stress tests, blood pressure, body mass index (BMI), and weight; (2) plasma markers associated with development of CAD such as lipids and triglycerides; and (3) molecular characteristics such as gene expression signatures and protein profiles.

B. To determine if patients with heart disease or risk factors that would promote heart disease can achieve and adhere to the goals of a lifestyle change program in a non-residential, out-patient setting.

ELIGIBILITY:
Inclusion Criteria: at least one known risk factor for cardiovascular disease:

* Family history of CAD (first degree relative)
* Physician-diagnosed diabetes or stroke
* Overweight (BMI/=25) or obese (BMI>/=30)
* Total cholesterol >/=200, documented history of hypercholesterolemia, or currently taking lipid lowering medications
* History of smoking
* HDL </=44 mg/dl
* LDL >/=130 mg/dl or documented history of hyperlipidemia
* Elevated triglycerides (>/=200 mg/dl)
* Hypertension (systolic blood pressure >/=130 mmHg, diastolic blood pressure >/=85 mmHg, documented diagnosis of hypertension, or currently taking antihypertensive medications)
* Diabetes (fasting glucose >/=100 mg/dl, physician diagnosis of diabetes/pre-diabetes, or currently taking anti-glycemic medications)
* Post traumatic stress disorder (PTSD) or at risk for PTSD
* Insomnia (five hours of sleep per night or less) or sleep apnea

Exclusion Criteria:

* Age <18 years of age
* Unstable coronary syndromes, refractory congestive heart failure, uncontrolled arrhythmia, or high-grade uncorrected cardiac conduction abnormalities
* Any contraindication to components to Program, such as physical disabilities precluding stretching and aerobic exercise or medical conditions that preclude consumption of foods essential to Program diet
* Inability or unwillingness to give consent
* Significant left main stenosis (>50%) or ejection fraction <35% with no revascularization
* History of substance abuse (including alcohol) without self-certification of abstinence for at least three months
* Non-ambulatory (bedridden) individuals

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2009-04; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | Baseline, 4-6 months, 1 year, 18 months, 2 years, 30 months, 3 years
  Change in BMI

SECONDARY OUTCOMES:
Blood Pressure | Baseline, 4-6 months, 1 year, 18 months, 2 years, 30 months, 3 years
  Change in systolic and diastolic BP
Blood Lipids | Baseline, 4-6 months, 1 year, 18 months, 2 years, 30 months, 3 years
  Change in HDL, LDL, total cholesterol, and triglycerides

OTHER OUTCOMES:
Exercise Capacity | Baseline, 4-6 months, 1 year, 18 months, 2 years, 30 months, 3 years
  Change in exercise capacity defined by Bruce score on an exercise treadmill test

CONTACTS AND LOCATIONS:
Overall Officials: Darrell L Ellsworth, PhD, Principal Investigator — Windber Research Institute
Locations (1):
- Windber Research Institute, Windber, Pennsylvania, United States

REFERENCES:
- See also: Windber Research Institute — http://www.wriwindber.org